CLINICAL TRIAL: NCT04233645
Title: Effect of Educational Video on Patient Adherence and Completeness of Intake and Voiding Diaries
Brief Title: Voiding Diary Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000026784
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The group will be given a standard scripted verbal and identical written instructions plus the study group will be shown a 5-minute educational video (available at https://youtu.be/rvYfDc-Yfus ) which depicts key components of entering data on the diary. Patients in this group will also have online access to the video when they are filling out their diaries.
  Interventions: Other: 5-minute educational video; Other: Usual Care
- Usual Care Group (Active Comparator): The group will be given a standard scripted verbal and identical written instructions as per usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: 5-minute educational video — The 5-minute educational video depicts key components of entering data on the diary. Patients in this group will also have online access to the video when they are filling out their diaries.
  Arms: Study Group
Other: Usual Care — The groups will be given a standard scripted verbal and identical written instructions as per usual care.

SUMMARY:
The aim of this study is to evaluate patient adherence and completeness of intake and voiding diaries. The secondary goal is to compare the satisfaction and understanding of patients of the intake and voiding trial diaries directions.

DETAILED DESCRIPTION:
This is a randomized prospective study. All women who need to complete an intake and voiding diary at the Yale Urogynecology outpatient facilities will be invited to participate. After completion of the consent process, they will be randomized to one of two groups. Both groups will have their voiding diaries analyzed by three blinded experts and will be graded on completeness of the information filled out. The mean grade obtained from this process and the return rate of the voiding diaries will be the primary outcomes. The secondary outcomes will include a brief patient questionnaire on their satisfaction of the instructions with the voiding diary. The primary and secondary outcomes will be evaluated between the groups to determine the effectiveness of the video intervention.

ELIGIBILITY:
Inclusion Criteria:

* Need for intake and voiding diary completion
* Deemed to required return visit or follow up
* Able to read and write English

Exclusion Criteria:

* Dementia
* Prisoners
* Pregnant Patients
* Medical and physical handicaps which may interfere with completion of intake and voiding diary
* Medical and physical handicaps with viewing or understanding of the educational video
* Illiterate patients
* Patients who cannot speak and understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Voiding Diary Grade | 3 days
  Voiding diaries will be evaluated by 3 blinded experts for completeness. The average of these 3 grades will be used to evaluate the intervention compared to the usual care group. Data entries can either be a void, leak, or fluid intake. Each data entry will be identified as either a leak, void, or fluid intake and then given a score based on completeness. Then these scores will be averaged with all the same type of entries per day and totaled, for a maximum total per day of 9. The maximum score is 9. A higher score means that the diary is determined to be more complete. The lowest score is 0, meaning the voiding diary was not complete. Each of the three days will then be averaged giving a final quality score for the returned voiding diary.
Return Rate of Voiding Diaries | 3 days
  The rate of return of voiding diaries will be compared between the 2 groups.

SECONDARY OUTCOMES:
Patient Satisfaction: questionnaire | 3 days
  A qualitative measure developed for the study will be used to assess the patient satisfaction. It consists of 4 questions, 1 Likert and 3 Yes/No questions. Each of these questions will be compared between the 2 groups. The questions are:
  1. I was satisfied with the instructions given to me about how to complete a bladder diary (likert).
  2. I understood the instructions about how to complete a bladder diary Yes/No
  3. I referred back to my written instructions after I left the office Yes/No.
  4. I referred to my video instructions after I left the office yes/ no

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States